CLINICAL TRIAL: NCT03745456
Title: Hemostasis Profile in Patients With Severe Subarachnoid Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Santiago R. Leal-Noval, Senior, Hospitales Universitarios Virgen del Rocío
Other Study IDs: HUVRocio
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Subarachnoid Hemorrhage; Platelet Dysfunction; Coagulation Disorder
Keywords: Rotational Thromboelstrometry
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hemostatic Disorders | interventions — Blood Specimen Collection; Platelet Aggregation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for coagulation profile (ROTEM and clotting tests) and platelet function (ROTEM platelet and PFA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subarachnoid Hemorrhage patients: Patients with severe subarachnoid hemorrhage (Hunt and Hess 4-5, Fisher 3-4) will be included initially in the first 6 hours after the onset of symptoms.
  Interventions: Diagnostic Test: Blood samples for ROTEM and platelet function.

INTERVENTIONS:
Diagnostic Test: Blood samples for ROTEM and platelet function. — Thormoboelastometry is based on the measurement of elasticity of blood by continuous graphical logging of the firmness of a blood clot during clot formation and subsequent fibrinolysis

SUMMARY:
Patients with severe subarachnoid hemorrhage (SAH) may present platelet and coagulation dysfunctions immediately after the stroke on admission at the hospital, and persisting up to 3-4 weeks after the onset. This study aimed to investigate the platelet function as assessed by impedance agregometry (ROTEM Platelet) and platelet adhesion (PFA), and the coagulation profile as assessed by ROTEM, over three evolutive times.

DETAILED DESCRIPTION:
Patients with severe subarachnoid hemorrhage (SAH) present platelet and coagulation dysfunctions immediately after the stroke, at least two weeks after the onset of SAH. These alterations have been implicated in the presentation of delayed cerebral ischemia (DCI), vasospasm, deep vein thrombosis (DVT) and long-term neurological deterioration. The temporal presentation of the platelet dysfunction and coagulation has not consistently been established, nor have they been assessed with tests for specific platelet receptors. Objective. Primary: To document the platelet function and coagulation, in constant and fixed periods after the stroke onset, in patients with severe SAH, Hunt and Hess 4-5, Fisher 4. Secondary: Relationship between the patterns of hemostasis and coagulation and the presence of vasospasm, DCI and DVT. Method. Prospective, cohort study that will include (calculated sample size) 50 patients with severe SAH, recruited in the first 6 hours after the onset of symptoms. Twenty healthy volunteers (already recruited) will constitute the control group. Platelet function will be studied by platelet count, von Willebrand factor level, platelet function assay (PFA-100), and platelet ROTEM for specific stimulation of platelet receptors (ARATEM, ADPTEM, TRAPTEM). The coagulation will be investigated by conventional coagulation study, ROTEM EXTEM, ROTEM FIBTEM and factor XIII. In the group with SAH, blood samples will be drawn into the first 6 hours after the onset of symptoms (t0), in the period of 8 - 10 days after the stroke (t1) - period of maximum incidence of TBI and DVT - and 14- 16 days after the stroke (t2) in order to evaluate the late degree of coagulation alterations. Baseline values (t0) will be compared between subjects with HSA and the control group (intersubjects comparisons.). On the other hand, significant changes of the hemostasis and coagulation values among the times t0, t1 and t2 in the HAS group, will be also investigated (intra-subjects comparisons). Additionally, the relationship between the hemostasis and coagulation values evaluated at any of the specified time and the clinical outcome, as assessed by the presence of DCI, vasospasm, DVT or neurological deterioration at 3 months of follow-up (mRs> 3), will be also investigated

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with severe subarachnoid hemorrhage (Hunt and Hess 4-5, Fisher 3-4) will be included initially in the first 6 hours after the onset of symptoms.

Exclusion Criteria:

1. Patient with known coagulopathy or with ingestion of antiplatelet drugs or anticoagulants in the 15 days prior to the presentation of symptoms.
2. Patients in whom there is no confirmed arteriovenous malformation.
3. The patient or authorized family member denies informed consent.
4. High risk of imminent death, evaluated by the doctor in charge of the patient.
5. Hemoglobin <100 g / L and / or platelet count <100,000 microL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe subarachnoid hemorrhage (Hunt and Hess 4-5, Fisher 3-4) in the first 6 hours after the onset of symptoms
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
ROTEM, ROTEM platelet and PFA variations in patients wit SAH. | 1 month.
  Document the platelet function (ROTEM platelet and PFA) and coagulation (ROTEM), in constant and fixed periods after the presentation of the stroke, in patients with severe SAH, defined by Hunt and Hess 4-5, Fisher 3-4.

SECONDARY OUTCOMES:
Secondary outcomes | 6 months
  Relationship between hemostasis and coagulation patterns and the presence of vasospasm, Late Cerebral Ischemia and Deep Venous Thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Santiago R Leal-Noval, MD, Principal Investigator — Medical staff of Neuro Critical Care
Locations (1):
- Hospital Universitario "Virgen del Rocío", Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided